CLINICAL TRIAL: NCT01268930
Title: Comparison of Hemostatic Matrix and Bipolar Coagulation in Surgical Treatment of Endometriomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Salih Taskin, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hemostaticmatrix
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-12

CONDITIONS: Ovarian Reserve; Endometrioma
Keywords: ovarian reserve; endometrioma excision; hemostatic matrix; bipolar electrocoagulation; thermal injury
MeSH Terms: conditions — Endometriosis | interventions — FloSeal Matrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bipolar coagulation (Active Comparator): In this arm, after the complete excision of ovarian endometrioma, ovarian hemostasis is provided by bipolar electrocoagulation.
  Interventions: Procedure: Bipolar electrocautery for ovarian hemostasis
- Hemostatic matrix (Active Comparator): In this arm, after complete excision of ovarian endometrioma, ovarian hemostasis is provided by hemostatic matrix.
  Interventions: Procedure: hemostatic matrix (FloSeal)

INTERVENTIONS:
Procedure: Bipolar electrocautery for ovarian hemostasis — after surgical excision of ovarian endometrioma with cyst wall, bipolar electrocoagulation is used to control of bleeding.
  Arms: Bipolar coagulation
Procedure: hemostatic matrix (FloSeal) — after surgical excision of ovarian endometrioma with cyst wall, hemostatic matrix is administered to the bed of cyst for 2-3 minutes to control of bleeding. Then, area is rinsed and hemostasis is checked.
  Arms: Hemostatic matrix

SUMMARY:
In this study, impacts of hemostatic matrix and bipolar electrocoagulation on ovarian reserve in women undergoing ovarian endometrioma excision are compared.

DETAILED DESCRIPTION:
Endometriosis is defined as the existence of endometrial tissue outside of the uterine cavity. Ovaries are the most common effected sites and the disease causes endometriotic cysts in the ovaries. The treatment of endometriomas is still highly controversial. It is well known that the ovarian reserve is compromised as a result of endometriomas. Even though a variety of medical agents can be used to treat endometriomas, when endometriomas cause pelvic pain or infertility especially when they are > 4cm in size, surgical treatment can be offered. Even though there is no standard surgical treatment removal of cyst wall is usually the preferred method. Aspiration of cyst fluid and coagulation of the cyst wall have been practiced, however are associated with more recurrences.

Nevertheless, the impact of surgical treatment on ovarian reserve has not been clarified. There are mainly two types of ovarian injury during surgical removal of endometriomas. First, there is risk that the healthy ovarian tissue can be removed along with the cyst wall. Second, there is risk of of thermal injury that occurs after cyst removal during hemostasis by electrocoagulation.

By this context, investigating an alternative method to electrocautery which causes less thermal injury to ovary would open a new strategy in the treatment of infertile patients with endometrioma.

A new method "hemostatic matrix" has been developed to provide hemostasis. Endometriomas can be treated without thermal injury to healthy ovarian tissue using this method compared to bipolar coagulation.

In the literature, there is no controlled randomized study compared hemostatic matrix and bipolar coagulation for impact on ovarian reserve after treatment ovarian endometriomas.

There are two main principles when treating endometriomas. First, recurrence should not occur, and the second is minimal ovarian injury.

On the backgrounds of this philosophy, it can be hypothesized that hemostatic matrix can cause less damage to ovarian tissue compared to classical bipolar coagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in reproductive ages
* Presence of ovarian endometrioma at least 4 centimeter in size

Exclusion Criteria:

* Previous ovarian surgery
* Pregnancy
* Lactation
* Diabetes Mellitus, thyroid or adrenal disorders, hyperprolactinemia
* History or suspicion of malignancy
* Use of oral contraceptive drug, GnRH agonist or antagonist, danazol and other drug relation with ovarian function in last 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
preoperative and at 1 and 3 months postoperatively ovarian reserve differences will be measured by serum anti mullerian hormone between two groups (hemostatic matrix and bipolar coagulation groups) | within preoperative 1 week, postoperative at 1 and 3 months
  Group 1: after excision of ovarian endometrioma with its wall hemostatic matrix is used to provide hemostasis in the bed of endometrioma.
  Group 2: after excision of ovarian endometrioma with its wall bipolar elektrocoagulation is used to provide hemostasis in the bed of endometrioma.
  At the end of study antimullerian hormone values as an indicator of ovarian reserve will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty Hospital, Ankara, Turkey (Türkiye)